CLINICAL TRIAL: NCT02920723
Title: Follow-up of the Patients Included in the EXESAS Study : Analysis of the Profit of the Physical Activity for the Control Group and of the Preservation of a Regular Physical Activity for the Group Initially Trained
Brief Title: Follow-up of the Patients Included in the EXESAS Study
Acronym: FOLLOW_EXESAS
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Centre Hospitalier Universitaire de Saint Etienne (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: 1608082; 2016-A00859-42 (Other: ANSM)
Record Dates: First submitted 2016-09-29; First posted 2016-09-30 (Estimated); Last update posted 2018-11-05 (Actual); Status verified 2018-11

CONDITIONS: Sleep Apnea Syndromes; Sleep Apnea, Obstructives
Keywords: Sleep Apnea Syndromes; Sleep Apnea, Obstructives; Training
MeSH Terms: conditions — Sleep Apnea Syndromes

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Training (Experimental): For the patients who were allocated in the control group in the EXESAS study. In this group, patients will perform 3 sessions of one hour per week of the "NeuroGyV" training program. It is a physical activity program with one session of Nordic walking, one session of "aquagym" and one session of gymnastic. Program lasts 9 months.
  Interventions: Other: Training
- Control (Other): For the patients who were allocated in the training group in the EXESAS study. In this group, patients will receive only diets and physical activity counselling
  Interventions: Other: Control

INTERVENTIONS:
Other: Training
  Other Names: NeuroGyV program
  Arms: Training
Other: Control
  Arms: Control

SUMMARY:
Sleep apnoea affects more than 20% of people over 65 years and is largely underdiagnosed. It does multiply tenfold the occurrence of vascular events, particularly stroke. While Continuous Positive Airway Pressure (CPAP) is currently the Gold standard treatment to prevent cerebrovascular and cardiovascular events, with a major clinical benefit, long term adherence to CPAP is a significant problem and search for alternative treatment is essential.

DETAILED DESCRIPTION:
In the previous EXESAS study (NCT02463890) the investigators compare evolution of Apnea Hypopnea Index (AHI) in an exercise trained group performed through in a national based non-profit organization (Fédération Française d'éducation Physique et de Gymnastique Volontaire (FFEPGV)) using a medical established program (NeuroGyV) during nine months against a control group receiving only standard dietetic and physical activity counseling.

The first partial observations of the study EXESAS seem encouraging in the term of 3 months of training. However, in the longer term, there is not a coverage in the treatment of the moderate Sleep Apnea: Obstructive Syndrome (SAOS). Thus they can logically expect that the possible therapeutic effect of the exercise is not maintained in the long term after the stop of the training.

This nex study suggests studying the profit of the exercise on sleep apneas for the patients who were initially in the control group in the EXESAS study and to observe if the preservation of a regular physical activity for the group which was trained in EXESAS study is associated with a preservation of the AHI after the additional year of follow-up without additional intervention

ELIGIBILITY:
Inclusion Criteria:

* Included in the previous EXESAS study
* Signature of consent

Exclusion Criteria:

* Patients being already treated for sleep apnea or clinical status (cardiovascular comorbidities) justifying an immediate initiation of CPAP
* Daytime sleepiness (ESS score > 10)
* Known respiratory or heart disease (or discovering during stress test) contraindicated exercise training
* Patients with Parkinson's disease
* AHI > 30

Ages: 40 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 79 (Actual)
Dates: Start 2016-09-01 (Actual); Primary Completion 2018-08-21 (Actual); Study Completion 2018-08-21 (Actual)

PRIMARY OUTCOMES:
the AHI (number of Apnea+Hypopnea per hour) through polysomnography assessment after twelve months of follow-up in the training and the control groups | 12 months
  Apnea-Hypopnea Index (AHI)

SECONDARY OUTCOMES:
Percentage of patients with AHI<15 through polysomnography assessment after twelve months of follow-up in the training and the control groups. | 12 months
Percentage of patients with AHI>30 through polysomnography assessment after twelve months of follow-up in the training and the control groups. | 12 months
Change in high frequency (HF) of spectral analysis of heart rate variability (parasympathetic index) at 12 months of follow-up in the 2 groups | 12 months
Maximal aerobic capacity (VO2Max) | 12 months
  Correlation between the change in VO2max during stress test, walking distance during 6 minutes and AHI in the two groups
Population Physical Activity questionnaire (POPAQ) | 12 months
  Correlation between the change in daily physical activity energy expenditure (estimated by the POPAQ questionnaire) and AHI in the two groups
Daily physical activity energy expenditure | 12 months
  Correlation between the daily physical activity energy expenditure (estimated directly by an actimetry sensor for 7 days) and AHI in the two groups
Epworth sleepiness Scale | 12 months
  Comparison of the variation of Epworth Sleepiness Scale (ESS) after 12 months follow-up for the two groups
Pittsburgh questionnaire | 12 months
  Comparison of the variation of Pittsburgh questionnaire after 12 months follow-up for the two groups
Berlin questionnaire | 12 months
  Comparison of the variation of Berlin questionnaire after 12 months follow-up for the two groups
Changes in blood pressure - Baroreflex | 12 months
  Measure of autonomic function (parasympathetic activity) - quantified via changes in blood pressure

CONTACTS AND LOCATIONS:
Overall Officials: Frederic ROCHE, MD - PhD, Principal Investigator — CHU de Saint-Etienne
Locations (1):
- CHU de Saint-Etienne, Saint-Etienne, France

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- See also: Website of the FFEPGV (in french) — http://www.sport-sante.fr/accueil/